CLINICAL TRIAL: NCT04554173
Title: An Appraisal of Minimal Invasive Surgery for Thoracic Child Neurogenic Tumour. A Multicentric Study
Brief Title: An Appraisal of Minimal Invasive Surgery for Thoracic Neurogenic Tumour
Acronym: DIUOP
Status: Completed | Type: Observational
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 20-HPNCL-01
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2021-08

CONDITIONS: Neurogenic Thoracic Tumors
Keywords: surgery; pediatric; surgical resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- surgical resection neurogenic tumors
  Interventions: Procedure: surgical resection neurogenic tumors

INTERVENTIONS:
Procedure: surgical resection neurogenic tumors — Patient who was treated for a thoracic neurogenic tumor by minimally invasive surgery

SUMMARY:
Mediastinal neurogenic tumors are relatively rare in children. Surgical resection is essential. Minimal invasive surgery is more and more used in pediatric population, but his evaluation for resection of thoracic neurogenic tumors is little studied.

Thoracotomy has specific long terms post operative complications. When compared to thoracotomy, thoracoscopy shows less operative blood loss, shorter duration of chest tube ans length of stay.

Recently, the indications of thoracoscopic approach have been assessed according to the presence or absence of image-defined risk factors (IDRF) at diagnosis and after preoperative chemotherapy in a monocentric retrospective study.

The investigators aimed to conduct a multicentric retrospective study to assess the role of thoracoscopy in neurogenic thoracic tumours according to the presence or absence of IDRF at diagnosis, the surgical complications and outcome.

DETAILED DESCRIPTION:
Mediastinal neurogenic tumors are relatively rare in children. Surgical resection is usually essential in there treatment. Minimal invasive surgery with video assisted thoracic surgery is more and more used in pediatric population, but his evaluation for resection of thoracic neurogenic tumors is little studied.

Thoracotomy has specific long terms post operative complications including scoliosis, shoulder elevation, winged scapula and asymmetric nipples. When compared to thoracotomy, thoracoscopy shows less operative blood loss, shorter duration of chest tube and length of stay.

Recently, the indications of thoracoscopic approach have been assessed according to the presence or absence of image-defined risk factors (IDRF) at diagnosis and after preoperative chemotherapy in a monocentric retrospective study. The authors concluded that thoracoscopy could be used for all paravertebral locations without IDRF except the IDRF of T9-T12 location and the presence of an intraspinal component but should be avoided for perivascular locations due to tight adherences of the tumour to the vessels and hence the risk of important bleeding.

The investigators aimed to conduct a multicentric retrospective study to assess the role of thoracoscopy in neurogenic thoracic tumours according to the presence or absence of IDRF at diagnosis, the surgical complications and outcome.

ELIGIBILITY:
Inclusion Criteria:

All children operated for neurogenic thoracic tumors with minimal invasive surgery

Exclusion Criteria:

-

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children operated for neurogenic thoracic tumors with minimal invasive surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Reason of failure of thoracoscopy | at inclusion
  counting of number of bleeding and surgical difficulties for a period of 30 days after surgery

SECONDARY OUTCOMES:
Post operative complications | at inclusion
  duration of hospitalization
Post operative complications number 2 | at inclusion
  Duration of chest tube

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Pédiatrique de Nice CHU Lenval, Nice, France